CLINICAL TRIAL: NCT03832062
Title: Value of Analysing Under-utilised Leftover Tissue (VauLT)
Acronym: VauLT
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Ventana Medical Systems (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCR 4838
Record Dates: First submitted 2019-01-24; First posted 2019-02-06 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The investigators will be collecting leftover formalin-fixed surgical tissue homogenate and FFPE tumour blocks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Leftover surgical tissue homogenization — Leftover surgical tissue homogenization

SUMMARY:
Intratumour heterogeneity is well recognized in multiple cancer types and ultimately leads to therapeutic resistance. It also limits the ability of small samples to represent the whole tumour, having implications for diagnosis, molecular analysis and understanding of the tumour immune microenvironment. By blending- 'homogenizing'- leftover tumour tissue in excess of that required for diagnosistic purposes, one may create a more representative sample for analysis.

DETAILED DESCRIPTION:
In order to establish the feasibility of homogenization as a potential companion diagnostic tool, our study aims to 1) evaluate how many surgical cases have left over tissue amenable to homogenization and 2) pilot homogenization across multiple tumour types. The molecular profile of the homogenate will be compared to that obtained from the diagnostic specimen using next generation sequencing techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Leftover formalin-fixed tissue (ie that would be otherwise discarded by histopathology) from cancer surgery.
2. Tissues for Research consent has been provided.
3. Patient age >18yo.
4. Minimum of 1 gram of residual tumour remaining in leftover surgical tissue
5. Minimum of 1 gram of normal tissue present.

Exclusion Criteria:

1. Advanced Practitioner in histological dissection deems tumour sample to be inadequate.
2. Leftover surgical tumour tissue greater than 20kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Leftover formalin-fixed tissue from cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of cases from surgical lists with tumour remains greater than 1g across 8 tumour groups | 24 Months
  Surgical lists will be generated providing cases of all surgeries containing excess tumour tissue. The tissue will be dissected and weighed to determine if tumour tissue available is greater than 1g

SECONDARY OUTCOMES:
Median time (in minutes) required for dissection of the leftover surgical tissue into tumour, tumour-adjacent and normal tissue | 24 Months
  The time taken to dissected will be documented by recording the start and stop times of the procedure and noting this on a source document
Median time (in minutes) required for the blending (actual homogenization) of each tissue type | 24 Months
  The time taken to homogenize will be documented by recording the start and stop times of the procedure and noting this on a source document
Difference in molecular profile between the diagnostic block and the homogenized sample. This will be measured by next generation sequencing techniques across the 8 primary tumour types | 24 Months
  The molecular profile of the diagnostic block will be determined by next generation sequencing and the same will be done with the homogenized sample. This will allow a comparison to be made between the two sample types and determine the difference in molecular profile between the two

CONTACTS AND LOCATIONS:
Overall Officials: Samra Turajlic, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided